CLINICAL TRIAL: NCT06996470
Title: The Relationship Between Cervical Endurance Time and Eye Gaze Dual Time in University Students
Brief Title: The Relationship Between Cervical Endurance Time and Eye Gaze
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Ahliyya Amman University (Other)
Responsible Party: Principal Investigator, Atef Nadier, Assistant professor of orthopedic physical therapy, Al-Ahliyya Amman University
Other Study IDs: 1979
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Endurance Time During Gazing
MeSH Terms: interventions — Vestibular Evoked Myogenic Potentials

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: - Cervical Vestibular-Evoked Myogenic Potential (cVEMP) along the Sternocleidomastoid — Endurance time during gazing

SUMMARY:
46 normal students will participate at the study; they will be randomly divided (male and female) into 2 groups (23 for each group) The study will be conducted in physical therapy lab and Speech and hearing center at Allied medical school.

ELIGIBILITY:
Inclusion Criteria:

* Normal students

Exclusion Criteria:

* subjects achieving less than 20 mmHg in the CCFT test
* Students with cervical pain within the last six months

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: normal students at university, level 3
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2025-09-28 (Estimated); Study Completion 2026-03-28 (Estimated)

PRIMARY OUTCOMES:
Endurance time during gazing | at base line
  measured by seconds
Endurance time without gazing gazing | at base line
  measured by seconds
Attention Span Scale for Students | at base line
  Questionnaire
Cervical Vestibular-Evoked Myogenic Potential (cVEMP) | at base line

IPD SHARING:
Plan to Share IPD: Undecided